CLINICAL TRIAL: NCT04717531
Title: Pyrotinib as Neoadjuvant Agent for Non-objective Response Patients of HER2-positive Early Breast Cancer Treated by Trastuzumab, Pertuzumab, and Chemotherapy (PYHOPE-BC-104): a Randomized, Controlled, Phase Ⅱ Trial
Brief Title: Pyrotinib as Neoadjuvant Agent for Non-objective Response HER2-positive Early Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PYHOPE-BC-104
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: neoadjuvant; pyrotinib; HER2-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Trastuzumab; Protons; pertuzumab; Docetaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): 2 cycles of pyrotinib and trastuzumab with docetaxel followed by 4 cycles of pyrotinib, epirubicin, and cyclophosphamide (THB*2-ECB*4). The cycles repeated every 21 days.
  Pyrotinib: 400mg, qd, po, day 1-21; Trastuzumab: 6 mg/kg, day 1; Docetaxel: 100 mg/m2, day 1; Epirubicin: 90 mg/m2, day 1; Cyclophosphamide: 600 mg/m2, day 1.
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab; Drug: Docetaxel; Drug: Epirubicin; Drug: Cyclophosphamide
- Cohort B (Active Comparator): 2 cycles of trastuzumab and pertuzumab with docetaxel followed by 4 cycles of epirubicin and cyclophosphamide (THP*2-EC*4). The cycles repeated every 21 days.
  Trastuzumab: 6 mg/kg, day 1; Pertuzumab: 420 mg, day 1; Docetaxel: 100 mg/m2, day 1; Epirubicin: 90mg/m2, day 1; Cyclophosphamide: 600 mg/m2, day 1.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pyrotinib — 400mg, qd, po, day 1-21
  Other Names: B
  Arms: Cohort A
Drug: Trastuzumab — 6 mg/kg, day 1
  Other Names: H
Drug: Pertuzumab — 420 mg, day 1
  Other Names: P
  Arms: Cohort B
Drug: Docetaxel — 100 mg/m2, day 1
  Other Names: T
Drug: Epirubicin — 90mg/m2, day 1
  Other Names: E
Drug: Cyclophosphamide — 600 mg/m2, day 1
  Other Names: C

SUMMARY:
The study assesses the efficacy of neoadjuvant treatment with pyrotinib and trastuzumab with chemotherapy, mainly pathological complete response (pCR) rates in the breast and axilla.

And also assesses side effects, event-free survival (EFS), disease-free survival (DFS), distant disease-free survival (DDFS), and objective response rates (ORR).

DETAILED DESCRIPTION:
Investigational Medical Products (IMPs) will be pyrotinib (B), trastuzumab (H), pertuzumab (P), docetaxel (T), epirubicin (E), and cyclophosphamide (C).

Magnetic resonance imaging (MRI) will be performed at baseline and 2 cycles after neoadjuvant therapy with trastuzumab, pertuzumab, and docetaxel (THP*2). Non-objective response patients will be randomly assigned (2:1) to receive 2 cycles of pyrotinib and trastuzumab with docetaxel followed by 4 cycles of pyrotinib and epirubicin plus cyclophosphamide (THB*2-ECB[epirubicine, cyclophosphamide, and pyrotinib]*4, cohort A), or 2 cycles of trastuzumab and pertuzumab with docetaxel followed by 4 cycles of epirubicin plus cyclophosphamide (THP*2-EC*4, cohort B).

During the neoadjuvant therapy, the side effects and all the events were recorded and analyzed. After surgery, the efficacy of pCR rate and ORR were analyzed. And long time follow-up will also be performed to analyze EFS, DFS, DDFS, and ORR.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients between 18-70 years old. 2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. 3. Histologically confirmed HER2 (human epidermal growth factor receptor-2)-positive invasive breast cancer.

4. Non-objective response after 2 cycles of THP as neoadjuvant treatment. 5. Known hormone receptor status. 6. Patient has adequate bone marrow, liver, and renal function:

1. Hematological: White blood cell (WBC) count > 3.5 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 90 x109/L, and hemoglobin ≥ 90 g/dL.
2. Hepatic function: total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (except for Gilbert's syndrome); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times ULN.
3. Renal function: serum creatinine and BUN ≤ 1.5 x ULN, or creatinine clearance ≥ 50 ml/min/1.73 m2 for patients with creatinine levels above institutional normal.

8. LVEF ≥50% measured by echocardiography. 9. Fertile patients must use effective contraception (barrier method - condoms, diaphragm - also in conjunction with spermicidal jelly, or total abstinence. Oral, injectable, or implant hormonal contraceptives are not allowed).

10. Negative serum pregnancy test, within 2-weeks (preferably 7 days) prior to randomization (For women of childbearing potential).

11. Signed informed consent form (ICF).

Exclusion Criteria:

1. Metastatic breast cancer;
2. Previous (less than 10 years) or current history of malignant neoplasms, except for curatively treated: Basal and squamous cell carcinoma of the skin; Carcinoma in situ of the cervix.
3. Patients with a prior malignancy diagnosed more than 10 years prior to randomization may enter the study. Patients must have been curatively treated with surgery alone. Radiation therapy or systemic therapy (chemotherapy or endocrine) are NOT permitted. Prior diagnoses of breast cancer or melanoma are excluded.
4. Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial;
5. Major surgical procedure or significant traumatic injury within 14 days prior to randomization or anticipation of the need for major surgery within the course of the study treatment.
6. Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension (≥180/110), unstable diabetes mellitus, dyspnoea at rest, or chronic therapy with oxygen;
7. Known hypersensitivity reaction to one of the investigational compounds or incorporated substances.
8. Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures during study treatment.
9. Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | up to 30 weeks
  Number of patients with pCR (no invasive breast cancer in the breast and axilla)

SECONDARY OUTCOMES:
Number of patients with grade >3 adverse events as a measure of safety and tolerability | up to 30 weeks
  To describe the safety of the various regimens toxicity is compared between the two arms.
Objective response rate (ORR) | up to 30 weeks
  ORR is defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Disease-free Survival (DFS) | Following surgery, every 12 months until Year 10
  DFS was defined as the time from surgery to the first date of breast cancer relapse, second primary tumor (including contralateral breast cancer), or death without documented prior relapse. Data will be reported when they are mature and available, likely when a median of 3 years follow up has been reached.
Event Free Survival (EFS) | From date of randomization until follow-up to 10 years
  EFS will be defined as the time from random assignment to documentation of the first of the following events: discontinuation of study therapy due to protocol-defined progression prior to surgery; local, regional, or distant recurrence of breast cancer following curative surgery; a new breast cancer; another new onset malignancy; or death as a result of any cause.
Distant-disease- free survival (DDFS) | From date of randomization until follow-up to 10 years
  DDFS is defined as the time period from randomization to the first event.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Zha, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China